CLINICAL TRIAL: NCT04203589
Title: The Effect of New Holistic Early Intervention Approach (Explorer Babies): a Randomized Controlled Study
Brief Title: Explorer Babies Early Intervention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Zubeyir Sari, Associate Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2017.729
Record Dates: First submitted 2019-11-21; First posted 2019-12-18 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Premature; Developmental Disability; Cerebral Palsy; Motor Disorders; Development, Infant
Keywords: Premature; Developmental Disability; Motor Disorder; Cerebral Palsy; Early Intervention; developmental Support
MeSH Terms: conditions — Premature Birth; Developmental Disabilities; Cerebral Palsy; Motor Disorders

STUDY DESIGN:
Intervention Model Description: A parallel randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Explorer Early Intervention Program (Experimental): The Explorer Early Intervention Program is used in this group.
  Interventions: Behavioral: The Explorer Baby Early Intervention Program
- Neurodevelopmental Therapy (Active Comparator): Neurodevelopmental therapy is used in these group by two experienced and certificated physiotherapist
  Interventions: Other: Neurodevelopmental Therapy

INTERVENTIONS:
Behavioral: The Explorer Baby Early Intervention Program — Centered based intervention, once or twice a month, 6 months follow up
  Other Names: Explorer Baby
  Arms: The Explorer Early Intervention Program
Other: Neurodevelopmental Therapy — Centered based intervention, once or twice a month, 6 months follow up
  Other Names: Bobath
  Arms: Neurodevelopmental Therapy

SUMMARY:
Premature babies have a high risk of adverse developmental outcomes. Early intervention approaches are applied to reduce these adverse outcomes or support of developmental delay. Early intervention approaches may vary depending on developmental priorities. While some early intervention methods can consider body structured findings such as posture, tonus, muscle power, others may consider coaching family, enrichment of the environment. The explorer baby program is developed based on the trial and error process. The program tries to find an answer to a unique question: "how trial behavior in infants can be increased and which behaviors of the infants should be supported to increase their trial process?" The Explorer baby program tries to increase exploratory motor behaviors to facilitate development. For this aim, the program tries to explain how a baby learns new skills such as rolling, sitting, babbling, playing peek a boo, etc. in all domains of development while the baby lives in their natural environment. This study aims to investigate the effect of the explorer baby early intervention program.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effect of Explorer Baby Early Intervention Program on explorative motor behaviors, motor, language, and cognitive skills. The study is designed as a randomized controlled trial in which infants and their families are randomly assigned to the intervention group (Explorer Baby) or control group (neurodevelopmental therapy), stratified by birth weeks and educational level of the mother.

There is no developmental support program as standard care in Turkey for premature babies. So that neither intervention nor the control group doesn't take any other support. There will be an average of six intervention sessions during the 6 months intervention period. The assessments will take before intervention (T0), after 3 months after T0 (T1) and after six months after T0 (T2), corrected age one (T3), corrected age two (T4).

Intervention: EXPLORatory motor behavior based Early Intervention Program (Explorer Baby) is a developmental support program for babies and their families. Parents visit the early intervention center with their babies in a variable frequency. The first step of the program is to build up interaction between therapists and parents; worries of parents for the development of their babies, knowledge about child development, knowledge about play behaviors, how babies learn new skills, age-specific requirements of babies, build up interaction with babies and family members, describing blocks for development.

The second step is setting the play in the natural environment working with the family; how do families describe the play? If families want to support the ability of their babies kicking, reaching, rolling, communicate, or social interaction how should they organize the playground? Showing families some examples of enrichment of playground for specific aims.

The third step is observing babies' reactions; how do families motivate their babies for play? How do families encourage their babies for self-starting explorative behaviors? How do parents support making the voice of the baby more if the play context is meaningful for creating a voice? The program doesn't give specific play homework to improve specific skills. The program tries to enrich parents' knowledge about the effect on the behavior of babies in meaningful situations.

The control Group: The control group will take neurodevelopmental therapy. Neurodevelopmental therapy is commonly accepted as traditional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Born before than 33 weeks

Exclusion Criteria:

* congenital malformations, all levels of asphyxia, intracranial hemorrhage, periventricular leukomalacia.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) | This tool will be used to assess the change between the three-time points. These time points are before therapy (T0), during therapy (T1 - 3 months after T0) and after therapy (T2 - 6 months after T0)
  The Bayley III is assessing "Cognitive, Receptive Language, Expressive Language, Fine Motor, Gross Motor". Bayley III has a raw score, scale score, composite score, and growth percentile score. All of these scores will be given in the study. But only, the growth percentage score will be discussed as both the subareas and the total score as the primary outcome. Because only the percentage of growth gives the baby's level of development exactly day by day. The percentile score is between 0 and 100. A higher score means improvement is better. The changes in the growth percentage in pre-test and post-test (T0-T1, T1-T2, T0-T2) will be examined in-group. Also, the growth percentage scores of two groups will be compared before, during and after the therapy (intergroup). This tool will be used to assess the change between the three-time points.

SECONDARY OUTCOMES:
Age and Stage Questionnaire 2 (ASQ-2) | This tool will be used to assess the change between the three-time points. These time points are before therapy (T0), during therapy (T1 - 3 months after T0) and after therapy (T2 - 6 months after T0)
  The Ages and Stages Questionnaire 2 (ASQ-2) is a widely used screening tool for infants and young children's development assessing development in five domains: Communication, Gross Motor, Fine Motor, Problem Solving and Personal Social. It is is originally a parent-completed questionnaire and it includes six questions for every developmental area. There are three options for the answer "Yes (10 points), Sometimes (5 points), No (0 points)". The raw score is between 0 to 60 points. High points mean better development. The study will use the raw score of all developmental areas. The age range of ASQ-2 is 3 months to 72 months meaning the ASQ-2 will not be used for children younger than 3 months. Post-tests (T1-T2) results will be used for discrimination (according to the parent's view) between children with developmental delays and developing typically in two groups.
Parent Stress Index-4-Short Form (PSI SF-4) | This tool will be used to assess the change between the three-time points. These time points are before therapy (T0), during therapy (T1 - 3 months after T0) and after therapy (T2 - 6 months after T0)
  The questionnaire is assessing "Parental Distress, Parent-Child Dysfunctional Interaction, Difficult Child" subheadings. High points are mean high-stress behaviour. The raw score is between 36 to 180 points. There are no cut scores in the Turkish version of PSI-4 SF. The changes in the raw scores in pre-test and post-test (T0-T1, T1-T2, T0-T2) will be examined in-group. Also, the raw scores of two groups will be compared before, during and after the therapy (intergroup). This tool will be used to assess the change between the three-time points.
Infant Movement Motivation Questionnaire | This tool will be used to assess the change between the three-time points. These time points are before therapy (T0), during therapy (T1 - 3 months after T0) and after therapy (T2 - 6 months after T0)
  The Questionnaire is assessing four subheadings with 27 items: "Activity, exploration, motivation, adaptability". There are no cut scores in these in the Turkish version of the questionnaire. High points mean better development. The raw score is between 27 to 135 points. The changes in the raw scores in pre-test and post-test (T0-T1, T1-T2, T0-T2) will be examined in-group. Also, the raw scores of two groups will be compared before, during and after the therapy (intergroup). This tool will be used to assess the change between the three-time points.

CONTACTS AND LOCATIONS:
Overall Officials: Zübeyir Sarı, PhD, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study will share the outcomes of statistics by using tables, figures.

REFERENCES:
- [Background] Babik I, Galloway JC, Lobo MA. Infants Born Preterm Demonstrate Impaired Exploration of Their Bodies and Surfaces Throughout the First 2 Years of Life. Phys Ther. 2017 Sep 1;97(9):915-925. doi: 10.1093/ptj/pzx064. PMID 28605484
- [Background] de Campos AC, Savelsbergh GJ, Rocha NA. What do we know about the atypical development of exploratory actions during infancy? Res Dev Disabil. 2012 Nov-Dec;33(6):2228-35. doi: 10.1016/j.ridd.2012.06.016. Epub 2012 Jul 21. PMID 22820063
- [Derived] Altunalan T, Sari Z, Dogan TD, Hacifazlioglu NE, Akman I, Altintas T, Uzer S, Akcakaya NH. Early developmental support for preterm infants based on exploratory behaviors: A parallel randomized controlled study. Brain Behav. 2023 Nov;13(11):e3266. doi: 10.1002/brb3.3266. Epub 2023 Oct 5. PMID 37798860